CLINICAL TRIAL: NCT04636606
Title: The Efficacy of the Myofunctional Therapy on Oral Dysphagia in Patients With Temporomandibular Disorders
Brief Title: Efficacy of the Myofunctional Therapy on Oral Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, PT, Msc, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/131
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Dysphagia, Oral Phase; Temporomandibular Disorders
Keywords: Oral Dysphagia; Temporomandibular Disorders; Quality of Life; Pain
MeSH Terms: conditions — Deglutition Disorders; Temporomandibular Joint Disorders; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home Exercise (Active Comparator): Home Exercise program includes educational training program about parafunctional activities of patients having oral dysphagia with temporomandibular disorders. Program includes stretching and strengthening of masticatory and neck muscles and posture exercises as well as diaphragmatic breathing exercises.
  Interventions: Procedure: Home Exercise
- Manual Therapy Combined with Home Exercise (Active Comparator): Manual Therapy includes deep friction massage and myofascial relaxation techniques to masticatory and neck muscles, active and resistant temporomandibular joint movements, temporomandibular joint distraction and mobilization, stretching techniques to the temporomandibular joint, mobilization of upper cervical joints.
  Home Exercise program includes educational training program about parafunctional activities of patients having oral dysphagia with temporomandibular disorders. Program includes stretching and strengthening of masticatory and neck muscles and posture exercises as well as diaphragmatic breathing exercises.
  Interventions: Procedure: Manual Therapy Combined with Home Exercise
- Orofacial Myofunctional Therapy combined with Manual Therapy and Home Exercise (Active Comparator): Orofacial Myofunctional therapy includes stretching the tongue muscles, tongue rotation exercises, isometric and isotonic strengthening of the tongue, special maneuver, effortful swallow exercise, strengthening exercise of hyoidal muscles.
  Manual Therapy includes deep friction massage and myofascial relaxation techniques to masticatory and neck muscles, active and resistant temporomandibular joint movements, temporomandibular joint distraction and mobilization, stretching techniques to the temporomandibular joint, mobilization of upper cervical joints.
  Home Exercise program includes educational training program about parafunctional activities of patients having oral dysphagia with temporomandibular disorders. Program includes stretching and strengthening of masticatory and neck muscles and posture exercises as well as diaphragmatic breathing exercises.
  Interventions: Procedure: Orofacial Myofunctional Therapy combined with Manual Therapy and Home Exercise

INTERVENTIONS:
Procedure: Home Exercise — Educational training program about oral dysphagia in patients with temporomandibular disorders.
  Arms: Home Exercise
Procedure: Manual Therapy Combined with Home Exercise — Manual therapy program combined with educational training program about oral dysphagia in patients with temporomandibular disorders.
  Arms: Manual Therapy Combined with Home Exercise
Procedure: Orofacial Myofunctional Therapy combined with Manual Therapy and Home Exercise — Orofacial Myofunctional Therapy program with combination of Manual therapy and educational training program about oral dysphagia in patients with temporomandibular disorders.
  Arms: Orofacial Myofunctional Therapy combined with Manual Therapy and Home Exercise

SUMMARY:
The aim of the study is to analyze the effects of orofacial myofunctional therapy (OMT) on oral dysphagia (OD) in patients with temporomandibular disorders (TMD).

DETAILED DESCRIPTION:
60 subjects with TMD, according to the Research Diagnostic Criteria, will be included in the study after voluntary consent form will be filled out. Subjects will randomly be divided into 3 groups according to the order.

Home Exercise (n=20) will be the Group 1, Home Exercise combined with Manual Therapy (n=20) will be the Group 2, and Orofacial Myofunctional Therapy combined with Home Exercise and MT treatment (n=20) will be the Group 3.

Group 1 will include educational training program about parafunctional activities of TMD disorders and active exercises for masticatory and neck muscles with 10 repetitions, 3 times a day, and for 10 weeks.

Group 2 will receive home exercise training program and manual therapy program which is planned to last 30 minutes; will be applied twice a week, for 10 weeks.

Group 3 will include stretching and strengthening of the tongue muscles, tongue rotation exercises, effortful swallowing, strengthen the hyoidal muscles, which is planned to last 40 minutes, will be applied twice a week, for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 65 years old
* Patients with diagnosis of Group Ia, Ib, IIa and and III according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD)
* Having pain ≥ 4 according to the Visual Analog Scale
* Having score ≥2 points on the Eating Assessment Tool-10 questionnaire
* Patients who had difficulty in water swallowing tests

Exclusion Criteria:

* Ages under 18 and over 65 years old
* Patients with a diagnosis of Group II b,c according to the RDC / TMD evaluation
* Diagnosis of psychiatric illness
* Patients with musculoskeletal problems in which systemic specific pathological conditions such as cervical and / or temporomandibular joint (TMJ) problem malignancy, fracture, rheumatoid disease is proven
* Patients who have undergone any surgery related to the cervical and/or TMJ
* Patients with facial paralysis
* Patients with swallowing difficulties due to the neurological disorders
* Patients who have received physical therapy associated with TMJ in less than 6 months
* Patients with cognitive deficits
* Participation rate lower than 80% of the program schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at 10 weeks and 6 months | Baseline, 10 weeks, 6 months
  Visual Analog Scale will be used where patients will be asked to rate their pain on a scale from 0 to 10 with 0 indicating no pain and 10 the maximum worst pain, at the baseline and the end of 10 weeks intervention and at the end 6 months from baseline.
Change from Baseline in Tongue strength and endurance at 10 weeks and 6 months | Baseline, 10 weeks, 6 months
  Tongue strength will be assessed by Iowa Oral Performance Instrument with the measurement of muscle strength by tongue muscle pressure.
  Tongue endurance will be measured with the Iowa Oral Performance Instrument by quantifying the length of time that a patient may maintain 50% of his or her maximum pressure.
Change from Baseline in Jaw Function limitation at 10 weeks and 6 months | Baseline, 10 weeks, 6 months
  Jaw function limitation will be measured by the Jaw Functional Limitation Scale-20 (JFLS-20) where the patients will be asked from 1 to 10 points per item (higher scores indicate worse jaw function). The JFLS-20 has 3 subscales: Mastication (6 items), Vertical Jaw Mobility (4 items), and Emotional and Verbal Expression (10 items).
Change from Baseline in Swallowing dysfunction at 10 weeks and 6 months | Baseline, 10 weeks, 6 months
  The first evaluation for swallowing dysfunction will be assessed with 100 ml water swallow test (WST). For the WST, we will be ask participants to consume 100ml of water in the shortest amount of time. Patients will be assessed to have failed the WST according to published criteria of, (1) coughing or choking post swallow, (2) having a wet voice quality post swallow, or (3) being unable to drink the whole amount of water. Furthermore, the swallowing speed will be evaluated as the amount of consumed water divided by the elapsed time.
  The second evaluation for swallowing dysfunction will be assessed with Eating Assessment Tool-10 (EAT-10) questionnaire. The EAT-10 is a self-administered, symptom-specific outcome assessment for swallowing dysfunction, demonstrating good consistency, reproducibility, and validity. It consists of 10 questions answered in a scale of 0 to 4 (0: no problem to 4: severe problem), with the higher scores indicating severe dysphagic symptoms.
Change from Baseline in Quality of life at 10 weeks and 6 months | Baseline, 10 weeks, 6 months
  The quality of life will be evaluated with Swallowing-related Quality of Life questionnaire (Swal-QoL). The SWAL-QoL is a dysphagia specific quality of life instrument consisting of 44 items (11 scales) assessing ten QOL domains: food selection, burden, mental health, social functioning, fear, eating duration, eating desire, communication, sleep, and fatigue. Sleep and fatigue contribute to general QOL, whereas the other domains are contributors to dysphagia-specific QOL. The total SWAL-QOL score includes 23 items from seven domains.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Umut Rehabilitation Center, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No